CLINICAL TRIAL: NCT05214716
Title: Single Center, Randomized, Open Label, Prospective Clinical Trial of BioFire FilmArray Assay for Antimicrobial Treatment of Hospital-acquired or Ventilator-associated Pneumonia in Intensive Care Units
Brief Title: FilmArray Pneumonia Panel for Antimicrobial Treatment of HAP/VAP in Intensive Care Units
Acronym: FilmArray
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Even if the study period was extended, it was expected that the target subjects would not be able to be registered, so the study was terminated early.
Sponsor: Kyungmin Huh (Other)
Responsible Party: Sponsor-Investigator, Kyungmin Huh, Assistant Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-11-103
Record Dates: First submitted 2021-12-30; First posted 2022-01-31 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Pneumonia, Ventilator-Associated; Pneumonia, Hospital Acquired; Critically Ill
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Respiratory specimens from the subjects are tested by the FilmArray Pneumonia panel and the results are reported via an electronic health record system. Treating physicians may adjust empirical antibiotic regimens with assistance from the guidelines formulated by the study investigators. Other microbiologic tests, including cultures, are performed as per routine practice.
  Interventions: Diagnostic Test: FilmArray Pneumonia panel
- Control (No Intervention): Microbiologic tests, including cultures, are performed as per routine practice. No intervention is made on the antimicrobial treatment in the control arm.

INTERVENTIONS:
Diagnostic Test: FilmArray Pneumonia panel — A rapid molecular diagnostic test designed to detect 27 bacterial and viral species and 6 major resistance genes from respiratory specimens.
  Arms: Intervention

SUMMARY:
Microbiologic diagnosis of pneumonia is often limited by a long turnaround time of cultures. This randomized trial aims to evaluate the impact of BioFire FilmArray Pneumonia panel on (1) the proportion of appropriate/optimal early antibiotic regimen and (2) the time to the administration of appropriate antibiotics in patients treated for hospital-acquired or ventilator-associated pneumonia (HAP/VAP) in ICU.

DETAILED DESCRIPTION:
The study subjects are adults treated for HAP/VAP in ICU, who should be enrolled within 24 hrs since the first administration of antibiotics. Informed consent are obtained from the subjects or their legal proxies. Due to the unique characteristics of ICU and the current COVID-19 pandemic, consent may be obtained via telephone when given by legal proxies; written consent should be obtained later. The subjects who meet the inclusion criteria are randomized into either intervention and control arms in 1:1 ratio. Respiratory specimens from the subjects in the intervention arm are tested with the FilmArray Pneumonia panel. Other routine microbiologic tests are performed for the subjects in both arms. The results are reported via electronic medical record, and the treating physicians may adjust antibiotic regimen with the assistance from the guidance formulated by the study investigators. No intervention is made on the antimicrobial treatment in the control arm. Primary outcomes are (1) the proportion of appropriate/optimal early antibiotic regimen and (2) the time to the administration of appropriate antibiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 years or older
2. Diagnosed with hospital-acquired or ventilator-associated pneumonia and being treated in an intensive care unit
3. Patient or his/her legal proxy agrees to participate and is able to provide informed consent

Exclusion Criteria:

1. Has been treated with antibiotic for HAP/VAP for 24 hr or longer
2. Requires antibiotic treatment for indications other than HAP/VAP
3. Bacteria has been isolated from respiratory specimens within 7 days prior to screening
4. Immunocompromised host whose major differential diagnosis includes Pneumocystis jirovecii or cytomegalovirus pneumonia
5. Expected to die within 2 days since screening due to underlying disease
6. Has an advance directive against mechanical ventilation or cardiopulmonary resuscitation
7. Does not want to participate or unable to provide consent
8. Determined to be unfit by the study investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
The proportion of appropriate/optimal early antibiotic regimen | within 24 hours
  * "Appropriate" antibiotics: agents active in vitro
  * "Optimal" antibiotics: appropriate AND not overly broad. Spectrums of antibiotics are categorized with the following hierarchy: colistin > carbapenem > piperacillin-tazobactam/4th generation cephalosporins > other beta-lactams/fluoroquinolones; for gram-positives, glycopeptides/linezolid > no glycopeptides/linezolid)
  * Early antibiotic regimen is defined as antibiotics administered ≤24 hr since the initiation of antibiotic treatment
The time to the administration of appropriate antibiotics | within 30 days
  time interval between the first dose of antibiotics and the first dose of antibiotics confirmed active in vitro

SECONDARY OUTCOMES:
30-day mortality (all-cause) | within 30 days
  death of any cause within 30 days since the initiation of antibiotic treatment
ICU mortality | within 30 days
  death of any cause while staying in the ICU within 30 days since the initiation of antibiotic treatment
Hospital and ICU length of stay | Through study completion, an average of 9 months
  length of hospital and ICU stay
Ventilator-free day | within 30 days
  the number of days that the patient was not on mechanical ventilation within 30 days since the initiation of antibiotic treatment
Dialysis-free day | within 30 days
  the number of days that the patient was not on hemodialysis (including continuous renal replacement therapy) within 30 days since the initiation of antibiotic treatment
Incidence of acute kidney injury | within 30 days
  Acute kidney injury is defined using the RIFLE (Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease) criteria.
Incidence of Clostridioides difficile infection | within 30 days
  C. difficile infection is defined as 3 or more defecations of unformed stool per day with a positive enzyme immunoassay or PCR for C. difficile toxin.
Acquisition of multi-drug resistance organism during hospital stay | within 30 days
  Multi-drug resistance (MDR) is defined as an in vitro resistance against 1 or more agents in 3 or more antibiotic classes. Methicillin (or oxacillin) resistance of Staphylococcus and vancomycin resistance of Enterococcus spp. are classified as MDR.
Duration of antibiotic treatment | within 30 days
  the number of days that the patient was administered with antibiotics for the treatment of pneumonia within 30 days since the initiation of antibiotic treatment
Total medical cost in the ICU | within 30 days
  total medical cost for the patient care in the ICU
Compliance to FilmArray guidance (intervention arm only) | within 30 days
  The proportion of early antibiotic regimens that complied with the recommendation in the guidance.

CONTACTS AND LOCATIONS:
Overall Officials: Kyungmin Huh, MD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No